CLINICAL TRIAL: NCT04701151
Title: Nordic Urothelial Cancer Research Group Study on Reduced BCG Dwell-Time in High Risk NMIBC
Brief Title: NORTH-REG Dwell-Time Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jørgen Bjerggaard Jensen (Other)
Collaborators: Aarhus University Hospital (Other); Herlev Hospital (Other); Odense University Hospital (Other); Aalborg University Hospital (Other); Regional Hospital West Jutland (Other); Rigshospitalet, Denmark (Other); Zealand University Hospital (Other); Landspitali University Hospital (Other); Sahlgrenska University Hospital (Other); Region Örebro County (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, Consultant, MD, DMSc Department of Clinical Medicine, Aarhus University, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-003112-27
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Side Effect of Drug
MeSH Terms: interventions — BCG Vaccine

STUDY DESIGN:
Intervention Model Description: multi-center, multi-national, two-armed, randomized, open-label, investigator-initiated clinical controlled - phase IV trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Study Subjects randomized to the interventional arm will be assigned to BCG induction therapy once-weekly for 6 weeks and subsequent 1 year of maintenance (6+3x3) of which dwell-time during the first of the 6 induction instillations is 2 hours.
  If side effects are registered before the second and all further instillations, Study Subject in the intervention arm will be reduced in dwell-time according to the grading of side effects as given by the study algorithm.
  Interventions: Drug: Bacillus Calmette Guerin
- Control (Active Comparator): The Study Subjects will be treated according to guidelines with BCG instillation therapy once weekly for 6 weeks and subsequent 1 year of maintenance therapy (6+3x3) with 2 hours of dwelltime.
  Interventions: Drug: Bacillus Calmette Guerin

INTERVENTIONS:
Drug: Bacillus Calmette Guerin — The same dose of the drug will be given in both arms but the dwell-time will be adjusted for the subjects in the intervention arm according to the grading of side effects given by the study algorithm.

SUMMARY:
Previous studies show that the majority NMIBC patients experience side effects to BCG and therefore terminate the instillations before completing all planned instillations. This will increase their risk of recurrence and potential cystectomy. The purpose of this study is to investigate if NMIBC patients who experience severe side effects to BCG instillations will experience fewer or less severe side effects if reducing dwell-time of BCG instillations.

The study will include patients from Denmark, Iceland, Norway and Sweden.

DETAILED DESCRIPTION:
Approximately 8,000 patients are diagnosed with bladder cancer (BC) in the Nordic countries every year. The majority of BC patients are diagnosed with non-muscle invasive bladder cancer (NMIBC). The majority of NMIBC are treated with Bacillus Calmette-Guérin vaccine (BCG) as adjuvant treatment but for carcinoma in situ it is the primary treatment. BCG is known to give a lot of side effects both local and systemic, the severity of these can lead to premature termination of the treatment.

The object of this PhD project is to investigate if reduced dwell time, the time the BCG is in the bladder, will decrease the severity of side effects due to BCG instillations.

This will be investigated in a Nordic setting and the project will be done as a two-armed randomized clinical trial.

By decreasing the severity of side effects, we hypothesize the number of patients completing all planned instillations will increase and thereby decrease the risk of the BC evolving into a more aggressive type.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at the time of signing the Informed Consent Form
* Signed Informed Consent Form
* Patients with NMIBC where BCG therapy including maintenance for 1 year is planned for one of the following histopathological findings:
* Ta high grade without CIS
* CIS with or without previous or concomitant Ta tumors
* T1 with or without CIS
* Is, according to the Investigator's judgement, able to comply with the trial protocol
* Ability to understand the Patient Information Sheet orally and in writing

Exclusion Criteria:

* Previous BCG instillations within the last 2 years, because of the risk of not having cleared potential previos side effects.
* T1 tumors where re-resection had not been performed
* TUR-B, bladder biopsy or traumatic catheterization within 2 weeks.
* Previous or current MIBC
* Progression defined as progrssion to T1-tumour, T2+_tumour or cystectomy irrespectievely of indication or development of metastatic urothelial cancer irrespectively of tumour stage
* Contraindications to BCG
* Incontinence
* Bilateral nephrostomy catheters; unilateral nephrostomy catheter is allowed if permanent for the duration of all inistallations with BCG and a normally functioning kidney.
* Need for catheter a demeure at the time of instillation
* Immune Suppressing medication (cancer therapy e.g cytostatic medicinal products, radiation, local and systemic steroids like e.g. prednisolone is permitted)
* Reduced immune response (leukaemia, lymphoma)
* Known allergy or sensitivity to BCG
* HIV infection
* Signs of active tuberculosis
* Any type of previosly radiation therapy involving the bladder.
* Concomitant invasive cancer within 5 years other than non-melanoma skin cancer and protate cancer without metastasis
* Current urinary tract infection
* Patient with visible hematuria
* Current alcohol and/or drug abuse
* Has a mental or legal incapacitation or another condition which impair the subject's ability to participate
* Has participated in another interventional clinical study and treatment with another investigational product 30 days prior to randomization
* For women study subjects: Pregnancy or breastfeeding
* For women Study subjects of childbearing potential: unless they are using highly effective methods of contraception from the first BCG instillations until 14 days after last dose of BCG treatment, which are defined as total abstinence, female sterilization, use of oral methods of contraception or placement of an intrauterine contraception devices.
* For male Study Subjects: unless they are using highly effective methods of contraception from the first BCG instillation until for 14 days after last dose of BCG treatment, which is defined as total abstinence or use of condoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Completion of instillations | 5 years
  Number of Study Subjects completing all 6 induction instillations and subsequent maintenance installations for 12 months (6 + 3 x 3)

SECONDARY OUTCOMES:
Recurrence rate | 5 years
  Recurrence rate within 24 months in Study Subjects with initial complete response

CONTACTS AND LOCATIONS:
Locations (11):
- Denmark (7):
  - Aarhus University Hospital, Aarhus, Aarhus N
  - Department of Urology, Aalborg University Hospital, Aalborg
  - Department of Urology, Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Regional Hospital Gødstrup, Herning
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde
- Landspitali University Hospital, Reykjavik, Iceland
- Sweden (3):
  - PO Sahlgrenska Universitetssjukhuset, Gothenburg
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No